CLINICAL TRIAL: NCT05305599
Title: Double-blind, Randomized, Placebo-controlled, Phase II Dose-finding Study Comparing Different Doses of ZED1227 Capsules With Placebo in the Treatment of Non-alcoholic Fatty Liver Disease (NAFLD) With Significant Fibrosis
Brief Title: Different Doses of ZED1227 vs. Placebo in NAFLD
Acronym: NormaliZED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEC-11/NAS
Record Dates: First submitted 2022-03-04; First posted 2022-03-31 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: NAFLD; Liver Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis | interventions — ZED1227

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ZED1227 (low dose) 10 mg (Experimental)
  Interventions: Drug: ZED1227
- ZED1227 (middle dose) 25 mg (Experimental)
  Interventions: Drug: ZED1227
- ZED1227 (high dose) 50 mg (Experimental)
  Interventions: Drug: ZED1227
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZED1227 — ZED1227 is a peptidomimetic designed to inhibit the activity of human tissue transglutaminase 2 (TG2).
  Arms: ZED1227 (high dose) 50 mg; ZED1227 (low dose) 10 mg; ZED1227 (middle dose) 25 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, multicenter, placebo-controlled, comparative, exploratory phase II dose-finding trial. The trial will be conducted with four treatment groups in the form of a parallel group comparison and will serve to compare oral treatment with daily doses of 20, 50, or 100 mg ZED1227 vs. placebo for the treatment of patients with NAFLD with fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Has provided signed informed consent
* Is a male or female ≥ 18 and < 75 years of age
* Has diagnosed NAFLD
* Has diagnosed significant fibrosis (stages 2 or 3)

Exclusion Criteria:

* Has a history of significant alcohol consumption (an average of > 20 g/d in females and > 30 g/d in males)
* Has a history or presence of any other significant concomitant liver diseases
* Has diagnosed type 1 diabetes mellitus (T1DM)
* Has presence of cirrhosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Relative change of PRO-C3 levels | 12 weeks
  Relative change (%) of serum levels of PRO-C3 between baseline and the EOT.

SECONDARY OUTCOMES:
Incidence of adverse events | from baseline to 16 weeks
  Incidence of treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, University Medical Centre, Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany